CLINICAL TRIAL: NCT06522178
Title: Anesthetic Techniques and Clinical Outcomes in the Oldest-old Patients Operated for Orthopedic Surgery: A Seven-year Retrospective Analysis of Data in a Third Level Hospital
Brief Title: Oldest-old Patients Anesthesia in Orthopedic Surgeries
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Ass-Prof, Istanbul Medeniyet University
Other Study IDs: Oldest-old Patient Anesthesia
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group I patients contained those who were between 80 (included) and 89 (included) years of age.
  Interventions: Other: Patient' ages
- Group 2: Those who were 90 years of age and above were included in Group II
  Interventions: Other: Patient' ages

INTERVENTIONS:
Other: Patient' ages — Patients were divided into two groups according to their ages.

SUMMARY:
Average life span, life expectancy, and the number of older people, aged 65 years and over, have increased during the last decades. As life expectancy increased, the rate of emergency and elective surgical interventions has also increased in the older age group. Although good health is required to reach an advanced age, over time, organ functions may deteriorate, and some challenges may develop that will negatively affect the balance of homeostasis. Stress, such as trauma or surgery, can cause deterioration in organ functions or aggravation of impaired functions. The risk of developing undesirable events is higher, due to the diminished reserve and function, during anesthesia applied to these patients. There is a limited number of studies in the literature about the relation between the anesthesia technique and morbidity and mortality in oldest old patients operated for orthopedic surgery. In this study, we aimed to analyze the data of the oldest-old patients operated on for orthopedic surgery between 2016-2022, retrospectively, and to investigate the relationship between anesthesia technique and adverse effects including morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Aged 80 years and above
* Underwent orthopedic surgery

Exclusion Criteria:

* Those who had the operation with local anesthesia

Ages: 80 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of 1356 oldest-old patients underwent orthopedic surgery between January 02 2016 and December 31 2022 in our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1356 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality | one month after operation
  postoperative mortality
Anesthesia Techniques | up to 6 hours
  Data were also analyzed and compared with groups and between groups according to the applied anesthesia technique (general anesthesia versus regional anesthesia).
Type of operation | up to 6 hours
  Orthopedic surgery type

SECONDARY OUTCOMES:
Presence and type of comorbidities | 6 month period before operation
  Hypertension, dementia, asthma, COPD (Chronic obstructive pulmonary disease), CHF (Chronic Heart Failure), CAD (Coronary artery disease), DM (Diabetes mellitus), valvular heart disease, history of pulmonary emboli, electrolyte imbalance, presence of cancer, renal diseases, history of cerebrovascular disease, endocrine diseases, neurologic diseases, other chronic diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided